CLINICAL TRIAL: NCT06077890
Title: Effectiveness of Digital Rehabilitation (SIMPLI.REHAB) in Hand Arthritis: A Randomized Clinical Trial
Brief Title: Effectiveness of Digital Rehabilitation (SIMPLI.REHAB) in Hand Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Responsible Party: Principal Investigator, Eugénio Moita Gonçalves, Principal Investigator, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 62/2023-1
Record Dates: First submitted 2023-09-24; First posted 2023-10-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Arthritis, Psoriatic; Arthritis, Rheumatoid; Deformity, Hand; Limitation, Mobility; Hand Arthritis; Hand Deformity
Keywords: Physical and Rehabilitation Medicine; Digital Technology; Occupational therapy; Hand; Rehabilitation
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid; Hand Deformities; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention Group (Experimental): This group incorporates the SIMPLI.REHAB digital tool as a complementary strategy for a rehabilitation program, including flexibility exercises and muscle strengthening, manual dexterity and motor coordination training, thermotherapy, and education on joint protection principles.
  Interventions: Other: Digital Rehabilitation
- Conventional Intervention Group (Active Comparator): This group follows a conventional rehabilitation program delivered in a more traditional, non-digital manner to serve as a comparison to assess the superiority of the experimental intervention using SIMPLI.REHAB digital tool.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Digital Rehabilitation — Participants in this arm will undergo an in-person rehabilitation program coordinated by a Physiatrist and will be able to access home-based rehabilitation strategies through dynamic content provided by SIMPLI.REHAB digital tool.
  Arms: Digital Intervention Group
Other: Conventional Rehabilitation — Participants in this arm will undergo an in-person rehabilitation program coordinated by a Physiatrist and will be given home-based strategies in a printed paper brochure.
  Arms: Conventional Intervention Group

SUMMARY:
This study investigates the effectiveness of SIMPLI.REHAB, a digital tool employed as an interface for administering occupational rehabilitation programs to patients diagnosed with Rheumatoid and Psoriatic Arthritis. Both of these conditions are inflammatory joint disorders capable of causing significant morphofunctional alterations in the hands, especially in their advanced stages. The introduction of digital technology emerges as a complementary tool when implementing rehabilitation programs.

Utilizing a prospective, longitudinal, single-blinded experimental study, 35 patients will be allocated into two groups: one receiving a complementary digital intervention through SIMPLI.REHAB and the other through a conventional rehabilitation program. Each group consists of six patients and the program spans seven weeks, focusing on therapeutic exercises, training in manual dexterity, and motor coordination, among other interventions, led by a Physiatrist.

The study intends to measure outcomes based on functionality scores, pain, disease activity, joint range, grip, pinch strength, and manual dexterity, both before and after each intervention, in order to ascertain the efficacy of integrating dynamic content through the digital tool SIMPLI.REHAB, as a supplementary resource in occupational rehabilitation programs. The potential limitations of the study include potential losses of follow-up and difficulties in assessing adherence to the digital tool precisely. Nonetheless, the digital tool aims to augment functional gains in rehabilitation programs by providing patients with accessible dynamic content of home-based strategies.

DETAILED DESCRIPTION:
Rheumatoid arthritis and psoriatic arthritis are inflammatory joint conditions that often affect the distal extremity of the upper limb responsible for manual functionality. If these conditions progress, they can lead to significant morphofunctional alterations. Occupational rehabilitation programs are essential for controlling and improving functional limitations. With the advent of the COVID-19 pandemic, various technologies have emerged that allow the implementation of rehabilitation programs in distinct manners. This study aims to assess the effectiveness of an occupational rehabilitation program using the digital tool SIMPLI.REHAB as an interface for administering home-based strategies to patients diagnosed with rheumatoid and psoriatic arthritis compared to a conventional rehabilitation program.

Using a prospective, longitudinal, single-blinded experimental study of superiority and randomized block design, 35 patients will be allocated to two intervention groups. An experimental intervention group will integrate an occupational rehabilitation program using the digital tool SIMPLI.REHAB for smartphones, compared to a group for a conventional rehabilitation program using a leaflet. Each group will consist of 6 patients and the program duration will be 7 weeks. This rehabilitation program, coordinated by a Physiatrist, includes classes for therapeutic exercises for flexibility and muscle strengthening, training in manual dexterity and motor coordination, thermotherapy, and patient education on joint protection principles conducted by the Occupational Therapy Team. The primary outcome to be assessed will be the functionality score with the Disabilities of the Arm, Shoulder, and Hand questionnaire. The surrogate endpoints will be pain (numerical pain scale), disease activity (DAS-28/DAPSA), joint range (digit-o-meter), grip and pinch strength (dynamometer), and assessment of manual dexterity (Moberg Pickup Test; 9-Hole Peg Test, and Kapandji's Pinches). The measurement of outcomes will be done before and after each intervention.

This study aims to assess the effectiveness of integrating a digital tool that provides dynamic content as a supplement to an occupational rehabilitation program, compared to the strategy traditionally used in patients with rheumatoid or psoriatic arthritis with morphofunctional alterations in the hand. Certain study limitations may relate to losses of follow-up during the rehabilitation program period and difficulty in precisely assessing adherence to the digital tool. However, this tool will allow patients to access dynamic content of home-based strategies that will enhance the functional gains obtained in a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

" Must be referred patients from the Rheumatology Service of CHVNG/E. " Age 18 or older. " Must have a clinical diagnosis of either rheumatoid arthritis or psoriatic arthritis by a Rheumatology specialist, as per the diagnostic criteria of the American College of Rheumatology.

" Must present pain, joint stiffness, joint instability, or osteoarticular deformities in the joints of the wrist, hand, and fingers.

" Must have a functional impact with a QuickDASH score > 31.5. " Must be capable of using the SIMPLI.REHAB app on a smartphone with internet connectivity.

" Must possess digital literacy allowing the use of the app. " Must have the ability to understand and provide informed consent.

Exclusion Criteria:

"Presence of other medical conditions that might interfere with participation or interpretation of results, such as: neoplasms, other systemic autoimmune diseases, diabetic polyneuropathy and/or uncontrolled diabetes " Having had local surgery on the joint of the wrist, hand, and fingers or a history of fracture in the last 6 months.

" History of intra-articular or intramuscular corticoanesthetic infiltration in the previous 4 weeks.

" Inability to perform hand exercises due to significant understanding, cognitive, or physical limitation.

" Participation in an occupational rehabilitation program during the study period or in the last 6 months.

" Severe hearing loss or visual impairment. " Undergoing other types of therapies or localized interventions in the hand and fingers during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) Score | Average of 7 weeks
  Hand functionality in basic and instrumental daily life activities, occupational and artistic or sports activities, through the score in the Disabilities of the Arm, Shoulder and Hand (DASH) 30-item questionnaire, calculated before and after the intervention.
  For each question, the patient rates on a 5-point Likert scale. The total score will range from 0 (no disability) to 100 (severe disability). It is a valid and reliable questionnaire (Pearson r > 0.70; ICC(2,1) = 0.96), with a minimal clinically important difference ranging between 10.83 and 15. (33, 37, 38).
QuickDASH Outcome Measure | Average of 7 weeks
  Shortened version of the DASH questionnaire which includes 11 items for clinical and functional evaluation of the upper limb. The QuickDASH questionnaire assesses an individual's ability to complete daily life activities, the ability to bear load, as well as the intensity of symptoms. It is also a valid and reliable questionnaire (Pearson r > 0.70; ICC(2,1) = 0.90), with the minimal clinically important difference ranging between 15.91 and 20.

SECONDARY OUTCOMES:
Number of Participants with New Osteoarticular Deformities | Average of 7 weeks
  Classification of osteoarticular deformities
Rate of Rescue Medications Usage | Average of 7 weeks
  Proportion of Pain-relief medications used
Number of Participants with Assistive Devices | Average of 7 weeks
  Determine the use of assistive devices and/or orthosis

OTHER OUTCOMES:
Numeric Pain Scale | Average of 7 weeks
  Score on the Numeric Pain Scale pre and post-intervention The Numeric Pain Scale is a unidimensional measurement instrument for pain intensity, frequently used in rheumatic diseases. The reliability of this scale is high (r = 0.96 to 0.95) with also high validity (r = 0.86 to 0.95). The minimal clinically significant difference is estimated at 1.1 points in patients with arthritis. (30, 31
Range of Motion | Average of 7 weeks
  Joint range of motion using a digit-o-meter pre and post-intervention
Muscular Strength | Average of 7 weeks
  Measurement of muscular strength using a pinch and palmar grip dynamometer pre and post-intervention.
  Dynamometry for objective assessment of pinch and palmar grip strength will allow for the evaluation of muscle strength in the hand and fingers.
  The minimal clinically important difference is estimated to be between 5 to 6 kgs.
Moberg Pickup Test Score | Average of 7 weeks
  Tool for objective assessment of manual dexterity and fine motor coordination pre and post-intervention.
9-Hole Peg Test Score | Average of 7 weeks
  Tool for objective assessment of manual dexterity and fine motor coordination pre and post-intervention.
Kapandji score | Average of 7 weeks
  Tool for objective assessment of manual dexterity and fine motor coordination pre and post-intervention.
Disease Activity Index for Rheumatoid Arthritis Patients (DAS-28) | Average of 7 weeks
  Score on Disease Activity Index pre and post-intervention for Rheumatoid Arthritis Patients.
  The DAS-28, or Disease Activity Score in 28 joints, is a measure commonly used to assess disease activity in patients with rheumatoid arthritis. It evaluates the number of swollen and tender joints out of a total of 28, the patient's global assessment of their health, and an acute phase reactant (usually the erythrocyte sedimentation rate or C-reactive protein level). The DAS-28 provides a score that falls into one of the following categories to represent the patient's disease activity:Remission: DAS-28 < 2.6; Low disease activity: DAS-28 between 2.6 and 3.2; Moderate disease activity: DAS-28 between 3.2 and 5.1; High disease activity: DAS-28 > 5.1
Disease Activity Index for Psoriatic Arthritis Patients (DAPSA) | Average of 7 weeks
  Score on Disease Activity Index pre and post-intervention for Psoriatic Arthritis Patients.
  DAPSA stands for Disease Activity index for PSoriatic Arthritis. It is a tool used to assess disease activity in patients with psoriatic arthritis. The score is calculated by summing the scores of the number of tender joints (68 joints are assessed), the number of swollen joints (66 joints are assessed), patient's assessment of pain, the patient's global disease activity and C-reactive protein (CRP) level (mg/dl). Low disease activity if DAPSA ≤ 15, moderate disease activity if DAPSA > 15 and ≤ 28 and, finally, high disease activity if DAPSA > 28.

CONTACTS AND LOCATIONS:
Overall Officials: Eugénio M Gonçalves, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.; Ana M Campolargo, MD, Study Director — Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Locations (1):
- Centro Hospitalar de Vila Nova de Gaia-Espinho, E.P.E., Porto, Vila Nova De Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No